CLINICAL TRIAL: NCT06243692
Title: Lacosamide Versus Topiramate in Migraine, a Ranodmized Trial
Brief Title: Lacosamide Versus Topiramate in Migraine
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, Dr., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000023988
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Migraine Disorders
Keywords: lacosamide; topiramate; migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Lacosamide; Topiramate

STUDY DESIGN:
Intervention Model Description: We will assess The number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The safety of treatment was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent statistician generated a blocked randomization sequence using computer-generated random numbers; participants received either lacosamide or topiramate from a specially trained and qualified nurse. We prepared Sequentially numbered opaque sealed envelopes and 600 labels for each drug labeled Drug A or B. According to the randomization chart, put them into envelopes numbered 1 to 600. Envelopes were attached to the patient's files. Patients were recruited sequentially and were given enrolment numbers starting from 1, which were mentioned on their files. Files with the same number as the patient enrolment number were opened and the patients were assigned to receive drugs A or B. Drug A included lacosamide, and Drug B included propranolol. The statistical analysis was performed by an independent statistician who did not know the treatment protocol of groups A or B.
  Both groups received open-label 500-1000mg acetaminophen during acute attack.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- lacosamide arm (Active Comparator): The arm will include 300 migraine patients diagnosed according to ICHD3-beta criteria. All patients will receive Lacosamide 50 mg twice daily and Acetaminophen 500-1000 mg only in acute migraine attacks for 3 months. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The safety of lacosamide was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
  Interventions: Drug: Lacosamide 50 MG
- Topiramate arm (Active Comparator): The arm will include 300 migraine patients diagnosed according to ICHD3-beta criteria. All patients will receive topiramate 100 mg daily and Acetaminophen 500-1000 mg only in acute migraine attacks for 3 months. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The safety of lacosamide was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
  Interventions: Drug: Topiramate 50Mg Tab

INTERVENTIONS:
Drug: Lacosamide 50 MG — The arm will include 300 migraine patients diagnosed according to ICHD3-beta criteria. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The safety of treatment was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
  Other Names: group A
  Arms: lacosamide arm
Drug: Topiramate 50Mg Tab — The arm will include 300 migraine patients diagnosed according to ICHD3-beta criteria. We will assess The change in migraine days per 28 days, the number of migraine days after three months of treatment, and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14). HIT-6 score reduction in each group after three months of treatment. The safety of treatment was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.
  Other Names: group B
  Arms: Topiramate arm

SUMMARY:
Investigators aim to compare the effect of lacosamide versus topiramate in migraine by assessing the absolute reduction in MMD in each group, the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency.

DETAILED DESCRIPTION:
Investigators will enroll 600 migraine patients who are diagnosed according to ICHD3-beta criteria in our study and will use a questionnaire to detect their demographic and clinical features (disease duration, attack frequency, and duration, pain intensity assessed by the visual analogic scale and we have two groups the first group will include 300 patients and will receive 50 mg lacosamide twice daily and Acetaminophen 500-1000 mg in acute attack, and the second group will receive topiramate100 mg per day and Acetaminophen 500-1000 mg in acute attack for at least three months. Investigators will assess The number of migraine days after three months of treatment and the percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency (14).. HIT-6 score reduction in each group after three months of treatment. The safety of lacosamide was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.

ELIGIBILITY:
Inclusion Criteria:

- Naive migraine patients, according to the International Classification of Headache Disorders 3rd edition, aged 10-55 years,

Exclusion Criteria:

- Patients with major neurological disorders such as ( epilepsy, ischemic or hemorrhagic stroke, multiple sclerosis, mitochondrial diseases, brain tumors, and patients with essential tremors.

Patients with major systemic diseases such as malignancy, collagen, liver, and renal diseases.

Patients with cardiovascular diseases like hypertension (systolic blood pressure of more than 130 and/or diastolic blood pressure of more than 85 mm/Hg on at least three different occasions, diabetes (fasting plasma glucose level >126 mg/dl and/or a casual plasma glucose >200 mg/dl and/or HbA1C more than 6.5.

patients with valvular and ischemic heart diseases, bradycardia or heart blocks, congestive heart failure patients who received prophylactic treatment for migraine, patients with any contraindications to drugs used in the study Patients with topiramate or lacosamide contraindications

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-02 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
The change in migraine days per 28 days | 28 days
  The investigators will assess the change in migraine days per 28 days in each group.

SECONDARY OUTCOMES:
The total number of migraine days after three months of treatment | 3 months
  The investigators will assess the total migraine days after three months of regular use of 50 mg lacosamide twice daily and Acetaminophen 500-1000 mg in acute attack or topiramate (100 mg daily) and Acetaminophen 500-1000 mg in acute attack alone.
The percentage of patients who achieved ≥ 50% reduction in the monthly migraine days frequency compared to the baseline frequency. | 3 months
  We will assess The percentage of patients who achieved ≥ 50% reduction in the monthly headache days frequency compared to the baseline frequency in each group
HIT-6 score absolute reduction in each group after three months of treatment | 3 months
  The investigators assessed the absolute reduction in HIT6 score, the Headache Impact Test-6 (HIT-6) assessed the burden of headache in each group; the HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress, the patient answers each of the six related questions using one of the following five responses: "never", "rarely", "sometimes", "very often," or "always." These responses are summed to produce a total HIT-6 score that ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent. It has four impact grades: little-to-no impact (HIT-6 score: 36-49), moderate impact (HIT-6 score: 50-55), substantial impact (HIT-6 score: 56-59), and severe impact (HIT-6 score: 60-78)
The safety of lacosamide was evaluated by monitoring treatment-emergent adverse events (TEAE) for three months. | 3 months
  The safety of treatment was evaluated by monitoring and documenting treatment-emergent adverse events (TEAE) in patients through regular follow-up procedures for three months.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed G. Zeinhom, MD, Study Director — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
All the data supporting this research's findings may be available from the principal investigator Mohamed G. Zeinhom upon reasonable request.

REFERENCES:
- [Result] Lipton RB, Scher AI, Kolodner K, Liberman J, Steiner TJ, Stewart WF. Migraine in the United States: epidemiology and patterns of health care use. Neurology. 2002 Mar 26;58(6):885-94. doi: 10.1212/wnl.58.6.885. PMID 11914403
- [Result] Lipton RB, Liberman JN, Kolodner KB, Bigal ME, Dowson A, Stewart WF. Migraine headache disability and health-related quality-of-life: a population-based case-control study from England. Cephalalgia. 2003 Jul;23(6):441-50. doi: 10.1046/j.1468-2982.2003.00546.x. PMID 12807523
- [Result] Mushet GR, Miller D, Clements B, Pait G, Gutterman DL. Impact of sumatriptan on workplace productivity, nonwork activities, and health-related quality of life among hospital employees with migraine. Headache. 1996 Mar;36(3):137-43. doi: 10.1046/j.1526-4610.1996.3603137.x. PMID 8984084
- [Derived] Zeinhom MG, Khalil MFE, Almoataz M, Youssif TYO, Daabis AMA, Refat HM, Ebied AAMK, Georgy SS, Akl AZO, Ismaiel M, Ahmed SI, Eissa HF, Ibrahem AIDM, Hassan AM, Elshafei M, Egila AAE, Ahmed SR. Lacosamide versus topiramate in episodic migraine: a randomized controlled double-blinded trial. Ther Adv Neurol Disord. 2025 Dec 9;18:17562864251396529. doi: 10.1177/17562864251396529. eCollection 2025. PMID 41384236